CLINICAL TRIAL: NCT04739306
Title: A Randomized, Active-Controlled, Double-Masked, Parallel-Group, Phase 3 Study to Compare Efficacy and Safety of CT-P42 in Comparison With Eylea in Patients With Diabetic Macular Edema
Brief Title: Study to Compare Efficacy and Safety of CT-P42 in Comparison With Eylea in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-P42 3.1
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Macular Edema (DME)
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CT-P42 (Experimental)
  Interventions: Biological: CT-P42
- Eylea (Active Comparator)
  Interventions: Biological: Eylea

INTERVENTIONS:
Biological: CT-P42 — 2mg/0.05 mL by Intravitreal injection
  Arms: CT-P42
Biological: Eylea — 2mg/0.05 mL by Intravitreal injection
  Arms: Eylea

SUMMARY:
This is a Randomized, Active-Controlled, Double-Masked, Parallel-Group, Phase 3 Study to Compare Efficacy and Safety of CT-P42 in comparison with Eylea in Patients with Diabetic Macular Edema

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥18 years.
* Patient with DME secondary to DM involving the center of the macula (defined as the Optical Coherence Tomography [OCT] central subfield) in the study eye.

Exclusion Criteria:

* Patient who has only one functional eye.
* Patient who currently has, or has a history (where indicated) of active proliferative diabetic retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- II. Ocna klinika SZU, F.D.Roosevelt Hospital, Banská Bystrica, Slovakia

REFERENCES:
- [Derived] Brown DM, Wolf S, Veselovsky M, Veith M, Papp A, Mange S, Mondal LK, Romanczak D, Janco L, Chauhan R, Romanowska-Dixon B, Eremina A, Dusova J, Sagong M, Kim S, Bae Y, Kim S, Bae Y, Son D, Kang H, Choi S, Stanga PE. Long-Term Efficacy and Safety of CT-P42 in Patients with Diabetic Macular Edema: 52-Week Results from a Phase 3 Randomized Clinical Trial. Ophthalmol Ther. 2025 Nov;14(11):2769-2783. doi: 10.1007/s40123-025-01197-w. Epub 2025 Aug 29. PMID 40879891

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who were randomly assigned to either group administrated study drug by intravitreal injection (IVT) via a sigle-dose vial every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
  After the Main Study period, a total of 31 subjects, regardless of the treatment group in Main Study Period, were enrolled in a 4-week open-label, single-arm Extension study. The subjects were administrated 2 mg/0.05mL of CT-P42 by pre-filled syringe IVT injection at Extension Week 0 (1 dose).
Groups:
- CT-P42 (Main Study Period): Subjects who were randomly assigned to CT-P42 group (2mg/0.05 mL) administrated by intravitreal injection via a single-dose vial every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
- Eylea (Main Study Period): Subjects who were randomly assigned to Eylea group (2mg/0.05 mL) administrated by intravitreal injection via a single-dose vial every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
Period: Main Study Period
Arm/Group | CT-P42 (Main Study Period) | Eylea (Main Study Period)
Started | 173 | 175
Completed | 153 | 153
Not Completed | 20 | 22
Not completed — Adverse Event | 6 | 7
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — War in Ukraine | 1 | 1
Period: CT-P42 PFS (Extension Study Period)
Arm/Group | CT-P42 (Main Study Period) | Eylea (Main Study Period)
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P42 | Eylea | Total
Number analyzed (Participants) | 173 | 175 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.6) | 62.9 (10.3) | 62.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 78 | 145
  Male | 106 | 97 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 166 | 165 | 331
  Unknown or Not Reported | 2 | 5 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 61 | 63 | 124
  White | 112 | 112 | 224
Region of Enrollment [Number; unit: participants]
  Czechia | 19 | 18 | 37
  Estonia | 1 | 1 | 2
  Hungary | 21 | 20 | 41
  India | 51 | 53 | 104
  Latvia | 9 | 5 | 14
  Lithuania | 0 | 1 | 1
  Poland | 19 | 21 | 40
  South Korea | 10 | 10 | 20
  Russia | 6 | 8 | 14
  Slovakia | 24 | 23 | 47
  Spain | 8 | 9 | 17
  Ukraine | 5 | 6 | 11
BCVA score at Baseline [Mean (Standard Deviation); unit: letters] — Baseline visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 73 to 34 (= Acuity of 20/40 to 20/200) in the study eye were included; a higher score represents better functioning.
  letters | 60.3 (9.7) | 60.4 (10.1) | 60.4 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 8
Description: Mean change from baseline in BCVA as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) letters at week 8.
  Subjects with a BCVA ETDRS letter score of 73 to 34 (= Acuity of 20/40 to 20/200) in the study eye at Screening and Day 1 were included. Visual acuity of the study eye was assessed using the ETDRS charts; a higher score represents better functioning.
Time Frame: Baseline and Week 8
Population: Full analysis set (FAS) consists of all subjects who are randomly assigned and received at least 1 full dose of study drug during the Main Study Period. Missing data were not imputed unless methods for handling missing data are specified.
Measure: Least Squares Mean (Standard Error); unit: letters
Groups:
- CT-P42: Subjects received Intravitreal injection of CT-P42 (2mg/0.05 mL), every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
- Eylea: Subjects received Intravitreal injection of Eylea (2mg/0.05 mL), every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
Arm/Group | CT-P42 | Eylea
Number analyzed (Participants) | 169 | 172
letters | 9.43 (0.798) | 8.85 (0.775)
Statistical Analysis 1: Comparison: CT-P42 vs Eylea; Test type: Equivalence — Predefined equivalence margin: -3 letters to +3 letters; ANCOVA; Analysis conducted for study eye. Primary endpoint as the dependent variable, treatment as a factor, baseline BCVA and country as covariates; Estimated difference in LS means = 0.58, 90% CI 2-sided [-0.52 to 1.67]

2. Secondary Outcome: Mean Change From Baseline in BCVA at Week 52
Description: Mean change from baseline in BCVA as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) letters at week 52.
Time Frame: Baseline and Week 52
Population: Full analysis set (subjects analysed at Week 52). Missing data were not imputed unless methods for handling missing data are specified.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | CT-P42 | Eylea
Number analyzed (Participants) | 156 | 156
letters | 12.1 (8.9) | 11.1 (9.9)

3. Secondary Outcome: Proportion of Subjects Who Gained ≥15 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52
Description: Proportion of subjects who gained ≥15 letters from baseline in BCVA, assessed in change from baseline in ETDRS letters over time
Time Frame: Baseline and Week 52
Population: Full analysis set. Missing data were not imputed unless methods for handling missing data are specified.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P42 | Eylea
Number analyzed (Participants) | 173 | 175
Participants | 60 | 52

4. Secondary Outcome: Proportion of Subjects With a ≥2-step Improvement From Baseline in the ETDRS DRSS (Diabetic Retinopathy Severity Score) as Assessed by FP (Fundus Photography) at Week 52
Description: The ETDRS DRSS score was grouped into 13 severity scores based on the ETDRS Severity Level.
  DR absent (level 10); Mild to moderate nonproliferative DR (levels 20, 35, and 43); Moderately severe/severe/Very Severe nonproliferative DR (levels 47, 53 and 53E); Inactive/Mild/moderate/high-risk/advanced proliferative DR (levels 60, 61, 65, 71,75, 81, and 85)
Time Frame: Baseline and Week 52
Population: Full analysis set. Missing data were not imputed unless methods for handling missing data are specified.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P42 | Eylea
Number analyzed (Participants) | 173 | 175
Participants | 41 | 38

5. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CST) at Week 52 as Assessed on Optical Coherence Tomography (OCT)
Description: The mean change from baseline in Central Subfieldl Thickness as determined by Spectral domain- Optical coherence tomography (SD-OCT)
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | CT-P42 | Eylea
Number analyzed (Participants) | 151 | 154
micrometer | -220.7 (147.1) | -191.2 (137.0)

ADVERSE EVENTS:
Time Frame: Main Study Period: From Week 0 to 52 Weeks, Extension Study Period: On or After Extension Week 0, assessed up to 4 weeks
Description: Safety analyses were performed in the safety population and was pre-specified to only report the most severe event if one or more events were occurred to the same subject.
  Note: One patient who was randomly assigned to the Eylea group was administered CT-P42 at the Week 40 visit. This patient grouped as CT-P42 group for the safety set for Main Study Period.
Groups:
- CT-P42 (Main Study Period): Subjects received Intravitreal injection of CT-P42 (2mg/0.05 mL), every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
- Eylea (Main Study Period): Subjects received Intravitreal injection of Eylea (2mg/0.05 mL), every 4 weeks for 5 doses, then every 8 weeks for 4 doses up to Week 48.
- CT-P42 (Extension Study Period): Subjects were administrated 2 mg/0.05mL of CT-P42 by intravitreal injection via a single-dose pre-filled syringe at Extension Week 0 (1 dose).
Arm/Group | CT-P42 (Main Study Period) | Eylea (Main Study Period) | CT-P42 (Extension Study Period)
All-Cause Mortality (participants affected / at risk) | 3/174 | 2/174 | 0/31
Serious Adverse Events (participants affected / at risk) | 19/174 | 17/174 | 0/31
Other Adverse Events (participants affected / at risk) | 64/174 | 71/174 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P42 (Main Study Period) (N=174) | Eylea (Main Study Period) (N=174) | CT-P42 (Extension Study Period) (N=31)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral end plate inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P42 (Main Study Period) (N=174) | Eylea (Main Study Period) (N=174) | CT-P42 (Extension Study Period) (N=31)
Cataract (Eye disorders) | 6 (6) | 4 (4) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 4 (5) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 4 (5) | 0 (0) — Study eye
Diabetic retinal oedema (Eye disorders) | 17 (18) | 23 (26) | 1 (1)
Posterior capsule opacification (Eye disorders) | 4 (5) | 3 (3) | 0 (0)
Visual acuity reduced (Eye disorders) | 5 (5) | 4 (4) | 0 (0)
Vitreous floaters (Eye disorders) | 3 (3) | 4 (4) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 4 (5) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 10 (10) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 6 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (11) | 4 (5) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 5 (5) | 1 (1)
Intraocular pressure increased (Investigations) | 3 (5) | 4 (9) | 0 (0)
Intraocular pressure increased (Investigations) | 3 (5) | 4 (8) | 0 (0) — Study eye
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 7 (7) | 7 (7) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 11 (12) | 16 (17) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT04739306/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT04739306/SAP_001.pdf